CLINICAL TRIAL: NCT06550427
Title: Early Assessment of Aggressive B-Cell Lymphoma Treatment Response and Prediction of Recurrence Using Phased Variant Analysis With Next-Generation Sequencing
Brief Title: Early Assessment of Lymphoma Treatment Response Using Phased Variant Analysis With Next-Generation Sequencing
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Attending physician, National Taiwan University Hospital
Other Study IDs: 202404016RINB
Record Dates: First submitted 2024-08-08; First posted 2024-08-13 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Lymphoma; Hodgkin Lymphoma; T-cell Lymphoma; Waldenstrom Macroglobulinaemia
Keywords: Lymphoma; NGS; Phased Variant; Early Response Assessment; Early Outcome
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Lymphoma, T-Cell; Waldenstrom Macroglobulinemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — paraffin-embedded tissue sections, bone marrow blood samples and peripheral blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- lymphoma: Pathology proven lymphoma
  Interventions: Diagnostic Test: ctDNA analyzed by phased variant

INTERVENTIONS:
Diagnostic Test: ctDNA analyzed by phased variant — this observational cohort study is to investigate the correlation between ctDNA analyzed by phased variant and the early outcome of the disease.

SUMMARY:
Lymphoma is a prevalent lymphoid malignancy globally and in Taiwan. Large B-cell lymphoma (LBCL) is the most common subtype of aggressive B-cell lymphoma. LBCL's aggressive nature manifests through extranodal involvement, severe symptoms, and relative refractoriness to therapies, leading to a 5-year overall survival rate of 60-70% across developed countries and poorer outcomes in high-risk patients with primary refractory disease. Chemoimmunotherapy remains the primary treatment for LBCL, requiring comprehensive assessment through clinical and imaging examinations, biomarkers, and molecular testing. Currently, computed tomography (CT) and positron emission tomography (PET) scans are the standard modalities for treatment response evaluation, though their radioactive nature calls for the development of safer alternatives. Circulating tumor DNA (ctDNA) analysis has emerged as a promising field, providing insights into tumor molecular characteristics, clinical status, and treatment response by analyzing DNA fragments released from tumor cells into the bloodstream. Dynamic monitoring of ctDNA during treatment can effectively gauge therapeutic efficacy-decreasing ctDNA concentrations suggest successful treatment, while increasing levels may indicate treatment failure or tumor recurrence. The detection of ctDNA has been much improved through advances in next-generation sequencing (NGS) technologies, particularly taking advantage of analyzing phased variants, consecutive gene mutations on the same chromosome, enhances the sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

* • Pathology proven lymphoma

  * Age ≥ 18 years old

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: pathology proven lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-08-09 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between ctDNA analyzed by phased variant and early outcome of lymphoma | From the date of enrollment, up to 24 months or date of death from any cause.
  The primary endpoint of this observational cohort study is to investigate the correlation between ctDNA analyzed by phased variant and the early outcome of aggressive B cell lymphoma

CONTACTS AND LOCATIONS:
Overall Officials: Tai-Chung Huang, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided